CLINICAL TRIAL: NCT05872802
Title: Effectiveness of a Proprioceptive Neuromuscular With One of Eccentric Exercise Plus Acute Electrostimulation in the Eccentric Exercise Plus Acute Electrostimulation on the Weight Bearing Weight Bearing Lunge, Lateral Step Down and Drop Jump Tests in Drop Jump Test, in Professional Paddle Tennis Players
Brief Title: Effectiveness of a Proprioceptive Neuromuscular Proprioceptive Neuromuscular Facilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15/05/2023
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Proprioceptive Neuromuscular Facilitation
Keywords: Proprioceptive neuromuscular facilitation;; Paddle tennis; Ankle dorsiflexion range; Eccentric exercise; Neuromuscular electrostimulation
MeSH Terms: interventions — Electric Stimulation; Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proprioceptive neuromuscular facilitation group. (Active Comparator): Proprioception protocol for ankle dorsiflexion.
  Interventions: Other: proprioceptive neuromuscular facilitation
- Eccentric exercises and electrical stimulation group. (Experimental): Eccentric exercises and strengthening currents for ankle dorsiflexion.
  Interventions: Other: eccentric exercises and electrical stimulation

INTERVENTIONS:
Other: eccentric exercises and electrical stimulation — Eccentric exercises and strengthening currents to improve ankle dorsiflexion in professional padel players.
  Arms: Eccentric exercises and electrical stimulation group.
Other: proprioceptive neuromuscular facilitation — proprioceptive neuromuscular facilitation to improve ankle dorsiflexion in professional padel players.
  Arms: proprioceptive neuromuscular facilitation group.

SUMMARY:
Introduction: Paddle tennis is a popular sport which can cause lower limb injuries due to impaired flexibility, such as ankle dorsiflexion. To improve this, methods such as proprioceptive neuromuscular facilitation (PNF), eccentric exercises and electrical stimulation (NMES) can be used. Objective: To compare the effectiveness of a PNF program with one of eccentric exercise plus NMES in the weight bearing lunge, lateral step down and drop jump test in amateur paddle tennis players. Methods: Pilot randomized clinical trial involving 20 male amateur paddle tennis players.

Participants were randomly divided into two groups of ten. One group received a PNF protocol, while the another group was given an Eccentric+ NMES exercise protocol. During the study, range of dorsal ankle flexion (ROMDf) was measured, as well as the vertical jump and lateral step down capacity of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Be a professional padel player.
* Be over 18 years of age.
* Sign the informed consent to participate in the study.
* Completion of the IPAQ physical activity questionnaire (Annex 1) to assess the level of physical activity of the participants and to ensure that they meet the physical activity level of the participants and to ensure that they meet the requirements for requirements for participation in the study.

Exclusion Criteria:

* Traumatic or musculoskeletal history that may affect the performance of the study exercises, as determined in the exercises of the study.
* A neurological history that may cause impairment in the performance of the exercises.
* Use of orthoses that may generate alterations in the result.
* Difficulty in performing exercises as determined by the Physical Activity Readiness Questionnaire (PAR-Q)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Vertical jump | 1 month
  The protocol for the drop jump test proposes different heights ranging from 20 to 100 cm.
  cm to 100 cm. In our study, there is a height of 25 cm to assess knee valgus, which is considered optimal according to the literature.
  knee valgus, which is considered optimal according to the literature. The athlete, once on the The athlete, once on the box, should place his hands on his hips and drop from the top of the bench, cushion the impact and, once in the jumping position, perform a maximum vertical jump.
range of flexion ankle dorsiflexion | 1 month
  using the weight bearing lunge test. Once the maximum distance has been reached, we perform the measurement with the clinometer application, we calibrate the the inclinometer at the verticality of your tibia, precisely at the proximal third and measure the range of motion of the ankle, not the position reached.

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge Velázquez Saornil, Ávila, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Osawa Y, Oguma Y. Effects of vibration on flexibility: a meta-analysis. J Musculoskelet Neuronal Interact. 2013 Dec;13(4):442-53. PMID 24292614
- [Background] Sams L, Langdown BL, Simons J, Vseteckova J. The Effect Of Percussive Therapy On Musculoskeletal Performance And Experiences Of Pain: A Systematic Literature Review. Int J Sports Phys Ther. 2023 Apr 1;18(2):309-327. doi: 10.26603/001c.73795. eCollection 2023. PMID 37020441
- [Result] Moreno-Perez V, Soler A, Ansa A, Lopez-Samanes A, Madruga-Parera M, Beato M, Romero-Rodriguez D. Acute and chronic effects of competition on ankle dorsiflexion ROM in professional football players. Eur J Sport Sci. 2020 Feb;20(1):51-60. doi: 10.1080/17461391.2019.1611930. Epub 2019 May 9. PMID 31072261
- [Result] Moreno-Perez V, Del Coso J, Raya-Gonzalez J, Nakamura FY, Castillo D. Effects of basketball match-play on ankle dorsiflexion range of motion and vertical jump performance in semi-professional players. J Sports Med Phys Fitness. 2020 Jan;60(1):110-118. doi: 10.23736/S0022-4707.19.09918-3. Epub 2019 Oct 16. PMID 31640316
- [Result] Rabin A, Kozol Z, Moran U, Efergan A, Geffen Y, Finestone AS. Factors associated with visually assessed quality of movement during a lateral step-down test among individuals with patellofemoral pain. J Orthop Sports Phys Ther. 2014 Dec;44(12):937-46. doi: 10.2519/jospt.2014.5507. Epub 2014 Oct 27. PMID 25347229
- [Result] Rabin A, Portnoy S, Kozol Z. The Association of Ankle Dorsiflexion Range of Motion With Hip and Knee Kinematics During the Lateral Step-down Test. J Orthop Sports Phys Ther. 2016 Nov;46(11):1002-1009. doi: 10.2519/jospt.2016.6621. Epub 2016 Sep 29. PMID 27686412
- [Result] Reiner M, Tilp M, Guilhem G, Morales-Artacho A, Nakamura M, Konrad A. Effects of a Single Proprioceptive Neuromuscular Facilitation Stretching Exercise With and Without Post-stretching Activation on the Muscle Function and Mechanical Properties of the Plantar Flexor Muscles. Front Physiol. 2021 Sep 14;12:732654. doi: 10.3389/fphys.2021.732654. eCollection 2021. PMID 34594241
- [Result] Wilczynski B, Zorena K, Slezak D. Dynamic Knee Valgus in Single-Leg Movement Tasks. Potentially Modifiable Factors and Exercise Training Options. A Literature Review. Int J Environ Res Public Health. 2020 Nov 6;17(21):8208. doi: 10.3390/ijerph17218208. PMID 33172101